CLINICAL TRIAL: NCT05749250
Title: Ultrasound Cavitation for Treatment of Non-healing Ulcers in Critical Limb Ischemia
Brief Title: Ultrasound Cavitation Therapy for CLI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Lindner, MD, Professor of Medicine, Cardiovascular Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR220344
Record Dates: First submitted 2022-10-25; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cavitation therapy (Experimental): Subjects treated with cavitation energy
  Interventions: Device: Acoustic cavitation of ultrasound enhancing agents
- Control (No Intervention): Control subjects not treated with cavitation energy

INTERVENTIONS:
Device: Acoustic cavitation of ultrasound enhancing agents — Cavitation therapy
  Arms: Cavitation therapy

SUMMARY:
In this study, we will explore how ultrasound exposure of ultrasound contrast agents, which produces beneficial shear-mediated bioeffects, can be used to treat patients with severe non-healing ulcers secondary to peripheral arterial disease (PAD). The primary outcome measure is whether ultrasound exposure to microbubble contrast agents in the inflow artery and at the wound site can accelerate wound healing. A secondary outcome measure is whether cavitation-related changes occur in tissue perfusion in the treated limb and wound measured by ultrasound perfusion imaging and skin flow.

ELIGIBILITY:
Inclusion Criteria:

* Known history of unilateral or bilateral PAD diagnosed by reduced ankle-brachial index (<0.9) or non-compressible vessels
* Diagnosis of CLI (Rutherford class IV-VI), and a non-healing ischemic ulcer defined as no change in the prior 3 months.

Exclusion Criteria:

* Major medical illness other than PAD affecting the limb (muscle disease, blood diseases that influence flow or rheology, severe heart failure [NYHA class IV]).
* Pregnant or lactating females
* Hypersensitivity to any ultrasound contrast agent or to polyethylene glycol (PEG, macrogol).
* Hemodynamic instability (hypotension with systolic BP <90 mm Hg, need for vasopressors).
* Expected amputation or revascularization procedure within the ensuing 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Wound dimensions | 18 days
  Area of non-healing ulcer

SECONDARY OUTCOMES:
Wound granulation | 18 days
  Area of granulation tissue of the ulcer
Tissue perfusion | 18 days
  Laser speckle perfusion imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No